CLINICAL TRIAL: NCT06887114
Title: Effects of Mulligan-Based Lumbar Mobilization on Trunk Position Sense, Balance, and Gait in Stroke Survivors: A Randomized Study
Brief Title: Can Lumbar Mulligan Mobilization Improve Gait, Balance, and Trunk Position Sense After Stroke?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mustafa Ertuğrul Yaşa, Assocc. Prof., Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14.03.2024/02-592
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Balance Impairments in Stroke Patients
Keywords: Stroke, Lumbar Mobilization, Mulligan, Balance, Trunk Position Sense and Gait.
MeSH Terms: conditions — Stroke | interventions — Exercise Therapy

STUDY DESIGN:
Masking Description: Single (Outcomes Assessor) single (outcomes assessor) single (outcomes assessor) the evaulation of the patients will be carried out by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Participants in this group will receive a combination of Mulligan Sustained Natural Apophyseal Glides (SNAGs) and conventional exercises.
  Interventions: Other: Experimental Group (Mulligan Mobilization + Conventional Therapy)
- Control Group (Active Comparator): Participants in this group will receive conventional physiotherapy exercises
  Interventions: Other: (Conventional Therapy Only)

INTERVENTIONS:
Other: Experimental Group (Mulligan Mobilization + Conventional Therapy) — Mulligan Sustained Natural Apophyseal Glides (SNAGs) applied to the lumbar spine, combined with conventional rehabilitation exercises (neuromuscular training, stretching, strengthening, and balance exercises).
  Other Names: SNAGs technique with conventional rehab; Lumbar SNAGs with rehabilitation exercises; Mulligan spine mobilization with physical therapy exercises; Lumbar mobilization and functional rehabilitation
  Arms: Study Group
Other: (Conventional Therapy Only) — Neuromuscular training, stretching, strengthening, balance exercises, and gait training performed without Mulligan mobilization.
  Other Names: Conventional Physiotherapy; Standard Rehabilitation Exercises; Traditional Physiotherapy Treatment; Conventional Exercise Program; Conventional Physiotherapy with Balance and Strengthening Exercises
  Arms: Control Group

SUMMARY:
Stroke is a pathology caused by disturbances in the brain's arterial circulation, leading to high morbidity rates. Individuals who experience a stroke often face neurological impairments such as motor, sensory, and cognitive dysfunctions, which negatively impact muscle strength, postural control, sensation, and gait, reducing their independence in daily activities. Balance deficits in stroke patients increase the risk of falls and contribute to a fear of falling. Improving balance control is a key goal in rehabilitation. The importance of the trunk in balance control and rehabilitation is well-established, as it plays a central role in maintaining stability. In individuals with restricted lumbar mobility, weakened trunk muscles and altered muscle activation can lead to a reduction in proprioception, hip strategy, and spinal stabilization, further impairing balance. Combining conventional exercise approaches with other rehabilitation techniques has been shown to yield more effective outcomes. This study aims to investigate the effects of Mulligan-based lumbar spine mobilization on balance, trunk position sense, and gait in individuals with stroke.

DETAILED DESCRIPTION:
Stroke is a high-morbidity condition caused by a disruption in the brain's arterial circulation, resulting in various neurological impairments, including motor, sensory, and cognitive deficits. These impairments lead to a decrease in the individual's ability to perform daily activities independently, as muscle strength, postural control, sensation, and gait are negatively affected. Stroke patients often face an increased risk of falls due to balance deficits, which can also contribute to a significant fear of falling. Thus, improving balance control is an essential therapeutic goal in stroke rehabilitation.

The trunk plays a pivotal role in balance control, and it should be the primary focus in rehabilitation programs. In individuals with restricted lumbar mobility, weakened trunk muscles or altered muscle activation patterns lead to decreased lumbar proprioception, impaired hip strategy, and reduced spinal stabilization, all of which contribute to balance difficulties. Recent studies suggest that combining conventional rehabilitation techniques with other interventions can provide more effective results.

In stroke rehabilitation, different mobilization techniques are increasingly being used. One such approach is the Mulligan Concept, which is commonly applied in musculoskeletal disorders, particularly in the treatment of knee, ankle, and shoulder problems in stroke patients. However, there has been limited research on the effectiveness of Mulligan-based lumbar spine mobilization in stroke patients. The Mulligan technique, particularly the Sustained Natural Apophyseal Glides (SNAG) technique, may help improve the individual's ability to move the body freely and enhance mobility and function, ultimately increasing confidence and reducing psychological barriers such as the fear of movement.

This study aims to evaluate the effectiveness of Mulligan-based lumbar mobilization in enhancing balance, trunk position sense, and gait in individuals with stroke. By assessing the impacts of this technique, the study seeks to contribute to the development of more effective rehabilitation strategies that can improve functional outcomes and quality of life for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following conditions to be eligible for the study:

  * Diagnosed with stroke by a neurologist.
  * Aged 30 to 65 years.
  * First-ever stroke (single episode).
  * Stroke duration between 6 to 24 months.
  * Score of ≤3 on the Modified Rankin Scale (mRS).
  * Score of ≥24 on the Mini-Mental State Examination (MMSE).

Exclusion Criteria:

* Participants will be excluded if they meet any of the following conditions:

  * History of musculoskeletal disorders affecting the spine (e.g., cancer, scoliosis, spondylolisthesis, rheumatoid arthritis, ankylosing spondylitis).
  * Previous lumbar spine surgery.
  * Presence of neurological conditions other than stroke (e.g., Parkinson's disease, multiple sclerosis).
  * Severe visual impairment affecting balance or walking.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Static Balance Assessment (Mini-BESTest) | Baseline and After 4 Weeks
  The Mini Balance Evaluation Systems Test (Mini-BESTest) assesses balance control, including anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. It consists of 14 items scored from 0 to 28, with higher scores indicating better balance.
Static Balance Assessment (ALDA Balance Device) | Baseline and After 4 Weeks
  The ALDA Balance Device uses a motion sensor placed at the L3-5 vertebrae to assess postural sway. It records movement data via a wireless system to analyze balance responses.
Dynamic Balance Assessment (Trunk Impairment Scale - TIS) | Baseline and After 4 Weeks
  The TIS assesses trunk control in stroke patients through three subcomponents: static sitting balance, dynamic sitting balance, and coordination. The scale consists of 17 items, with a total score ranging from 0 to 23, where higher scores indicate better trunk control.
Dynamic Balance Assessment (Functional Reach Test - FRT) | Baseline and After 4 Weeks
  The Functional Reach Test evaluates balance stability by measuring the maximum distance a participant can reach forward while maintaining a fixed base of support. Three trials are conducted, and the average distance is recorded. A reach distance of 15 cm or less indicates a high fall risk.
Gait Performance (Dynamic Gait Index (DGI)) | Baseline and After 4 Weeks
  Assesses functional mobility and dynamic walking ability under different conditions (e.g., changing speeds, stepping over obstacles).
Gait Performance (10-Meter Walk Test) | Baseline and After 4 Weeks
  Measures gait speed by recording the time taken to walk 10 meters.
Trunk Position Sense (Proprioception) inclinometers test | Baseline and After 4 Weeks
  Inclinometers are among the most commonly used methods for measuring trunk position sense and proprioception. the participant will be guided into a 30° lumbar flexion position three times while standing and will be asked to memorize this position. Then, the participant will be instructed to close their eyes and attempt to replicate the same position. After returning to an upright stance, they will be asked to find the 30° flexion position again. This process will be repeated three times, and the results will be recorded.

SECONDARY OUTCOMES:
Fall Risk (Timed Up and Go (TUG) Test) | Baseline and After 4 Weeks
  Evaluates functional mobility by measuring the time taken to stand from a chair, walk 3 meters, turn, walk back, and sit down.
Cognitive Function (Standardized Mini Mental Test (SMMT)) | Baseline and After 4 Weeks
  Assesses cognitive status, including memory, attention, and visuospatial abilities.
Functional Independence (Barthel Index) | Baseline and After 4 Weeks
  Assesses independence in daily living activities such as mobility, self-care, and transfers.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Indivudual participant data will be available to the responsible researcher.